CLINICAL TRIAL: NCT00225823
Title: A Randomised, Double-Blind, Placebo-Controlled, Parallel Group, Multicentre Two Week Study to Evaluate the Efficacy and Safety of Once-Daily, Intranasal Administration of GW685698X Aqueous Nasal Spray 100mcg in Adult and Adolescent Subjects With Seasonal Allergic Rhinitis in Europe
Brief Title: Study In Adults And Adolescents With Seasonal Allergic Rhinitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFR103184
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Seasonal Allergic Rhinitis Intranasal Corticosteroid
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW685698X

SUMMARY:
Compare the efficacy and safety of an investigational nasal spray compared with placebo nasal spray in the treatment of seasonal allergic rhinitis. Allergic rhinitis is an inflammatory disorder of the upper airway that occurs following allergen exposure. The focus of this study, seasonal allergic rhinitis (SAR), is one type of allergic rhinitis that is triggered by the pollen from trees, grasses, and weeds. Commonly referred to as 'hay fever', it is characterized by sneezing, nasal congestion and pruritus, rhinorrhea, and pruritic, watery, red eyes.

ELIGIBILITY:
Inclusion criteria:

* Informed consent.
* Must be an outpatient.
* Females must be using appropriate contraception.
* Must have diagnosis of seasonal allergic rhinitis, adequate exposure to allergen.
* Must be able to comply with study procedures.
* Must be literate.

Exclusion criteria:

* A significant concomitant medical condition.
* Use of corticosteroids or allergy or medications or tobacco.
* Clinically significant abnormal ECG.
* Laboratory abnormality.
* Positive pregnancy test.
* Allergy to any component of the investigational product.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2005-05; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline over the entire treatment period in daily, reflective, total nasal symptom scores (rTNSS).

SECONDARY OUTCOMES:
Mean change from baseline over the entire tx period in AM, pre-dose iTNS. Mean change from baseline over the entire treatment period in rTOSS. Overall evaluation of response to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Latvia (2):
  - GSK Investigational Site, Liepāja
  - GSK Investigational Site, Riga
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Šiauliai
  - GSK Investigational Site, Vilnius
- Netherlands (6):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Arnhem
  - GSK Investigational Site, Assen
  - GSK Investigational Site, Leeuwarden
  - GSK Investigational Site, Schiedam
  - GSK Investigational Site, Tilburg
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Volgograd
- Sweden (4):
  - GSK Investigational Site, Ängelholm
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Västerås

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: FFR103184 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFR103184 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFR103184 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR103184 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFR103184 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR103184 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR103184 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register